CLINICAL TRIAL: NCT01468805
Title: Childhood Asthma Reduction Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110230; 11-E-0230
Record Dates: First submitted 2011-09-10; First posted 2011-11-10 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2013-11-15

CONDITIONS: Asthma
Keywords: Environmental Intervention; Indoor Allergens; Cockroach; Health Disparities; Multi-Center; Asthma; Environment
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Procedure: Cockroach mitigation/extermination

SUMMARY:
Background:

- Cockroach allergies are an important risk factor for asthma in inner-city households, especially in children. A new method for killing cockroaches may help children who live in households that have high numbers of cockroaches. Because most public health treatments target more than just cockroaches, this method could lower the costs of treating childhood allergies and asthma by focusing on the most likely source of the allergy.

Objectives:

- To test a new cockroach-killing method designed to reduce asthma in children exposed to cockroaches.

Eligibility:

* Children 5 to 14 years of age who have moderate to severe asthma.
* Children must live in a household that has a high number of cockroaches.

Design:

* Participants will be screened with a phone call and an initial home visit.
* Study doctors will place cockroach traps, and return after 3 days to check the number of roaches caught and killed. Dust samples will be collected from the house.
* Participants will have blood and lung function tests, and will be tested for allergies (including cockroach allergies).
* Some households will be treated for cockroaches at regular intervals, or more frequently if required by the study doctors.
* Participants will have regular checkup visits in their homes at months 1, 3, 6, 9, and 12 and short phone call interviews at months 2, 4, 6, 8 and 10 to study their asthma symptoms. The home visits will also check the cockroach levels in the house.

DETAILED DESCRIPTION:
Asthma is the most prevalent chronic childhood condition and is the most frequent cause of hospitalization among children. There are about 6.7 million children in the U.S. who currently have asthma, and nearly two of every three of these children had at least one attack in the past 12 months. Evidence suggests that exposure to cockroach allergen might be the most important risk factor for asthma in inner-city households. An environmental intervention targeting only cockroach allergen could potentially provide cost savings in a public health program over high cost multi-component interventions, if it could be shown to reduce asthma morbidity.

The primary objective of the Childhood Asthma REduction Study (CARES) is to evaluate the effectiveness of a novel cockroach eradication method, shown in prior studies to drastically decrease cockroach allergen levels, in reducing asthma morbidity in children with moderate to severe asthma who are both allergic and exposed to cockroach allergen. Additionally, the study will characterize relationships between cockroach infestation and other environmental allergen exposures, and asthma morbidity, as well as consider dynamic relationships between cockroach counts and observed allergen reductions over time; and use study data to identify mechanisms such as cleaning behaviors that may influence those relationships.

These objectives will be addressed through a prospective, randomized controlled, multi-site intervention trial in which 414 eligible children age 5 to 14 years who live in households with a confirmed trap count of 30 or more cockroaches over a 3-day period, are randomly assigned to one of two treatment groups. Treatment will be implemented at multiple intervals in the homes of children assigned to the intervention group. Children in both the intervention and control groups will receive clinical evaluations for asthma, home assessments of allergen exposures, educational materials on allergen exposures and asthma, and information on study results. Following 12-months of active data collection, the extermination treatment will be made available to the homes of children in the control group. The target sample size is 372 participants completing the study, equally divided into the two arms. Home environmental assessments following the enrollment visit will take place at enrollment, 1, 3, 6, 9, and 12 months. Clinical assessments will also be conducted in the home at enrollment and the 12-month visit. Primary outcome data will be collected during scheduled follow up phone calls every two months.

ELIGIBILITY:
* INCLUSION CRITERIA:

A child will be included in this study if the following criteria apply:

(Assessed during phone screening)

* Aged 5 to 14 years of age
* Physician diagnosis of asthma for at least one year prior to prescreening
* Parent/guardian able and willing to provide consent; child able and willing to provide assent
* Primary caretaker and child are able to speak English or Spanish
* Moderate to severe asthma as defined by the child experiencing one of the following:

  * One overnight hospitalization for asthma within the past 6 months,

OR

--Two unscheduled clinic or emergency department visits for asthma within the past 12 months

-Sleeps in the target home greater than or equal to 5 nights per week

(Assessed at beginning of enrollment/baseline visit)

* Target home has greater than or equal to 30 cockroaches trapped in a 3 day period
* Positive ImmunoCAP Rapid test result to cockroach allergen

EXCLUSION CRITERIA:

A child will be excluded from this study if the following criteria apply, as determined in the screening phone call and/or confirmed at the baseline visit:

* The child has other serious medical or chronic illnesses, other than asthma, such as:

  * Any hematologic, metabolic/endocrine, respiratory (other than asthma), cardiac or neurologic disorder requiring daily medications;
  * Any severe behavioral problem that prohibits the child or the child s caregiver from answering questions or following instructions;
  * Any autoimmune disease including rheumatoid arthritis, lupus, and myositis;
  * Any immune deficiency;
  * Any other serious medical condition such as juvenile diabetes mellitus, hypothyroidism, hyperthyroidism, cerebral palsy, hyperimmunoglobulin E syndrome, or diagnosed allergic bronchopulmonary aspergillosis.
* Plans to move within the 12 months of study enrollment
* Has no caregiver with access to a phone

Sibling or other household member currently participating in the study.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-09-04; Primary Completion 2013-11-15 (Actual); Study Completion 2013-11-15 (Actual)

PRIMARY OUTCOMES:
Change in the mean number of maximum asthma symptom days.

SECONDARY OUTCOMES:
Asthma-related medical care resource utilization, Lung function, Medication use, Cockroach Number and Allergen Reductions.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C Zeldin, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)